CLINICAL TRIAL: NCT05637840
Title: Longitudinal Study of Metabolic Content of Human Urine
Brief Title: Study of Metabolic Content of Urine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Morgridge Institute for Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-1111; A537700 (Other: UW Madison); SMPH/BIOMOLEC CHEM/BIOMOL CHM (Other: UW Madison); Protocol Version 9/28/22 (Other: UW Madison)
Record Dates: First submitted 2022-11-22; First posted 2022-12-05 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Metabolic Content of Urine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep limited (Experimental): Participants will be asked to limit their sleep
  Interventions: Other: Urine sample; Other: Sleep restriction
- No sleep limitation (Experimental): Participants will be asked to get their normal amount of sleep.
  Interventions: Other: Urine sample

INTERVENTIONS:
Other: Urine sample — Collection of 36-84 urine samples over a 14 consecutive day period.
Other: Sleep restriction — Participants will be asked to limit their sleep to 4 hours within a 24-hour period for 2 days in a row.
  Arms: Sleep limited

SUMMARY:
The purpose of this research study is to test the different components in urine and see if they can be matched to food, exercise and sleep that participants report. The researchers are trying to find out if urine would allow them to predict medical problems as they are happening. Participants are healthy volunteers who are willing to give urine samples on a daily basis, and can expect to be in the study for 28 days.

DETAILED DESCRIPTION:
The purpose of this research study is to analyze urine samples using Mass Spectrometry to identify metabolites that have the potential to be used for medical diagnosis. This data, along with data from wearable devices, will be combined and analyzed to correlate what an individual does on a daily basis with how their body metabolizes their choices. This type of data may provide insights into the origins and progression of diseases in a short time span.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Be able to provide informed consent
* Stated willingness to comply with all study procedures and have availability for the duration of the study

Exclusion Criteria:

* Presence of a condition(s) or diagnosis, either physical or psychological, that limits the ability to urinate in the collection apparatus
* Individuals who do not consistently get at least 6 hours of sleep per night
* Individuals who have a sleep disorder diagnosis.
* Individuals who live in the state of New York

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-11-18 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
Change in inflammation | Baseline to day 14
  Changes in inflammation will be measured by hs-CRP via short-term sleep restriction.
Correlate biohealth data with concentrations of urine metabolites | Daily for 14 days
  To explore connections between urine metabolite concentrations and others measures of health and lifestyle, biometric data will be collected using a FitBit watch (sleep and exercise), nutritional data (food logs) and a questionnaire (tobacco use). Urine will be analyzed using mass spectrometry to isolate metabolites. The metabolites will then be cross-referenced against databases of known metabolites in order to identify them and their disease associations.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Coon, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT05637840/ICF_000.pdf